CLINICAL TRIAL: NCT03080571
Title: To Evaluate the Safety, Feasibility and Clinical Outcome of Intraarterial Infusion of Bone Marrow Derived Mononuclear Cells in Subacute Ischaemic Stroke Patients
Brief Title: Intraarterial Stem Cells in Subacute Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Vikas Bhatia, Principal investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGIMER RADIOLOGY
Record Dates: First submitted 2017-03-07; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Ischemic Stroke; MCA Infarction
MeSH Terms: conditions — Ischemic Stroke; Infarction, Middle Cerebral Artery | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: test group :Stem cell plus standard care control group : standard care
Who Masked: Outcomes Assessor
Masking Description: PROBE design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stem cell group (Experimental): autologous BMMNC stem cells with standard care
  Interventions: Biological: autologous BMMNC stem cells; Other: standard care
- Control (Active Comparator): Patients randomised in this group received standard care only
  Interventions: Other: standard care

INTERVENTIONS:
Biological: autologous BMMNC stem cells — Autologous BMMNC injected in the ipsilateral MCA
  Arms: Stem cell group
Other: standard care

SUMMARY:
Stroke is a leading cause of morbidity and mortality.Acute ischemia causes irreversible damage to neurons and glial cells, leading to functional deficits and chronic sequelae with variable degrees of spontaneous recovery of function. Stem cells have been shown to enhance recovery through multiple immunomodulatory effects, neoangiogenesis and neurogenesis.

We conducted a prospective randomised end observer blinded study to evaluate primarily the safety of intraarterial autologous stem cells delivered to ipsilateral middle cerebral artery in acute and subacute stroke patients (0-15 days post ictus).Secondarily we aimed to evaluate the outcome on the basis of clinical evaluation and follow up imaging

DETAILED DESCRIPTION:
1. This study was done over a period of one and a half years from July 2015 to December 2016. A total of 229 patients who presented with acute middle cerebral artery stroke and admitted at Post graduate institute of medical education and research were evaluated for recruitment into this study.
2. Participants who satisfied the inclusion criteria were randomized at 1 week into control and stem cell infusion test group within 15 days of stroke onset.
3. Investigators evaluated 20 patients, with 10 each in control and stem cell infusion test group.
4. Participants in the test group were infused autologous bone marrow mononuclear cells through intraarterial route using a microcatheter which was placed in proximal ipsilateral M1 segment of MCA. Participants in the control group did not receive stem cell therapy. Rest of the pharmacological treatment and physiotherapy were similar in both groups for the period of 6 months.

5,Participants were evaluated with clinical and radiological follow up at 6 months.

ELIGIBILITY:
Inclusion Criteria: Requires presence of all of the following

1. Age range 20-80 years symptoms
2. Signs of clinically definite MCA stroke (0 to 14 days post ictus)
3. National Institute of Health Stroke Scale (NIHSS)> 7,
4. Stroke clinically and on imaging conforming to the MCA territory,
5. Recanalization/patency of involved M1 segment of MCA on imaging
6. Patency of carotid arteries for intra-arterial access of cerebral circulation

Exclusion Criteria: Requires presence of any of the following

1. cerebral hemorrhage on CT/MRI
2. Imaging evidence of M1-MCA segment complete occlusion
3. Hemodynamic instability
4. Known defect of clotting or platelet function
5. Severe co-morbidity precluding intra-arterial intervention
6. Hepatic or renal dysfunction
7. Pregnant patients
8. Patient likely to be unavailable for follow-up
9. Patients with evidence of chronic illness or advanced cancer
10. Patient already dependent in activities of daily living before the present acute stroke i.e. pre stroke mRS >3
11. Refusal to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in National Institutes of Health Stroke Scale | 6 month
  increase in National Institutes of Health Stroke Scale more than / equal to 4 points
symptomatic intracranial hemorrhage | 6 month
new ischemic lesion | 6 month
Death | 6 month

SECONDARY OUTCOMES:
modified rankin score | 6 months
  A modified rankin score of 0-1 in patients with National Institutes of Health Stroke Scale of 8-14 at the admission and modified rankin score of 0-2 in patients with National Institutes of Health Stroke Scale >14 at the admission.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Gupta, DM, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh; Vikas Bhatia, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moniche F, Gonzalez A, Gonzalez-Marcos JR, Carmona M, Pinero P, Espigado I, Garcia-Solis D, Cayuela A, Montaner J, Boada C, Rosell A, Jimenez MD, Mayol A, Gil-Peralta A. Intra-arterial bone marrow mononuclear cells in ischemic stroke: a pilot clinical trial. Stroke. 2012 Aug;43(8):2242-4. doi: 10.1161/STROKEAHA.112.659409. Epub 2012 Jul 3. PMID 22764211
- [Background] Battistella V, de Freitas GR, da Fonseca LM, Mercante D, Gutfilen B, Goldenberg RC, Dias JV, Kasai-Brunswick TH, Wajnberg E, Rosado-de-Castro PH, Alves-Leon SV, Mendez-Otero R, Andre C. Safety of autologous bone marrow mononuclear cell transplantation in patients with nonacute ischemic stroke. Regen Med. 2011 Jan;6(1):45-52. doi: 10.2217/rme.10.97. PMID 21175286
- [Background] Suarez-Monteagudo C, Hernandez-Ramirez P, Alvarez-Gonzalez L, Garcia-Maeso I, de la Cuetara-Bernal K, Castillo-Diaz L, Bringas-Vega ML, Martinez-Aching G, Morales-Chacon LM, Baez-Martin MM, Sanchez-Catasus C, Carballo-Barreda M, Rodriguez-Rojas R, Gomez-Fernandez L, Alberti-Amador E, Macias-Abraham C, Balea ED, Rosales LC, Del Valle Perez L, Ferrer BB, Gonzalez RM, Bergado JA. Autologous bone marrow stem cell neurotransplantation in stroke patients. An open study. Restor Neurol Neurosci. 2009;27(3):151-61. doi: 10.3233/RNN-2009-0483. PMID 19531871
- [Background] Savitz SI, Misra V, Kasam M, Juneja H, Cox CS Jr, Alderman S, Aisiku I, Kar S, Gee A, Grotta JC. Intravenous autologous bone marrow mononuclear cells for ischemic stroke. Ann Neurol. 2011 Jul;70(1):59-69. doi: 10.1002/ana.22458. PMID 21786299
- [Background] Friedrich MA, Martins MP, Araujo MD, Klamt C, Vedolin L, Garicochea B, Raupp EF, Sartori El Ammar J, Machado DC, Costa JC, Nogueira RG, Rosado-de-Castro PH, Mendez-Otero R, Freitas GR. Intra-arterial infusion of autologous bone marrow mononuclear cells in patients with moderate to severe middle cerebral artery acute ischemic stroke. Cell Transplant. 2012;21 Suppl 1:S13-21. doi: 10.3727/096368912x612512. PMID 22507676